CLINICAL TRIAL: NCT00004879
Title: An Open Label, Multiple Dose, Dose-Rising Clinical Trial of the Safety of ABX-EGF in Patients With Renal, Prostate, Pancreatic, Non-Small-Cell Lung, Colorectal, or Esophageal Cancer
Brief Title: Monoclonal Antibody ABX-EGF in Treating Patients With Renal (Kidney), Prostate, Pancreatic, Non-Small Cell Lung, Colon or Rectal, Esophageal, or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067539; UCLA-9906078; ABX-EG-9901; UCLA-9906078-04B; NCI-G00-1673
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Kidney Cancer; Lung Cancer; Pancreatic Cancer; Prostate Cancer
Keywords: recurrent renal cell cancer; recurrent prostate cancer; recurrent colon cancer; recurrent rectal cancer; recurrent non-small cell lung cancer; recurrent pancreatic cancer; recurrent esophageal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Kidney Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Carcinoma, Renal Cell; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Panitumumab

INTERVENTIONS:
Biological: panitumumab

SUMMARY:
RATIONALE: Monoclonal antibodies such as ABX-EGF can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody ABX-EGF in treating patients who have either renal (kidney), prostate, pancreatic, non-small cell lung, colon, rectal, esophageal, or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of monoclonal antibody ABX-EGF in patients with renal, prostate, pancreatic, non-small cell lung, colorectal, esophageal, or gastroesophageal junction cancer.
* Determine the pharmacokinetics and the dose-response relationship of this drug in this patient population.
* Evaluate the clinical effect of this drug in this patient population.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive monoclonal antibody ABX-EGF IV over 1 hour once weekly on weeks 0-3* (enrollment for the weekly dosing schedule completed as of 4/21/03 [with the exception of patients undergoing full pharmacokinetic analyses, described below]) OR once every 2 weeks on weeks 0, 2, 4, and 6* OR once every 3 weeks on weeks 0, 3, 6, and 9*. Patients undergoing full pharmacokinetic analyses receive a loading dose on week 0 and the subsequent 3 doses on weeks 3-5.

NOTE: *All patients receive a total of 4 doses.

Cohorts of 2-8 patients receive escalating doses of monoclonal antibody ABX-EGF until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 or 3 patients experience dose-limiting toxicity.

Patients are followed every 2 weeks for 5 weeks.

PROJECTED ACCRUAL: A total of 76 patients will be accrued for this study within approximately 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Renal cell cancer (RCC)

    * Prior nephrectomy required
  * Prostate cancer

    * Failed prior primary therapy (e.g., surgery, radiotherapy, or chemotherapy)
    * Failed prior hormonal therapy (e.g., antiandrogen, luteinizing hormone-releasing hormone inhibitor, or orchiectomy)
  * Pancreatic cancer

    * Failed at least 1 prior standard therapy regimen for unresectable metastatic disease
  * Non-small cell lung cancer

    * Failed at least 1 prior standard therapy regimen for unresectable metastatic disease
  * Colorectal cancer

    * Received 1 or more prior chemotherapy regimen(s) for advanced metastatic disease
  * Esophageal cancer

    * Failed prior primary therapy (e.g., surgery, radiotherapy, or chemotherapy)
  * Gastroesophageal junction cancer
* Evaluable disease
* Epidermal growth factor receptor overexpression

  * Tumor tissue must yield the sum of 1+, 2+, or 3+ staining in at least 10% of evaluated tumor cells
* No uncontrolled brain metastases
* No evidence of disease progression or regression after a 30-day washout period

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100% OR
* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* AST/ALT no greater than 2 times upper limit of normal (ULN) (3 times ULN for liver metastases)
* Alkaline phosphatase no greater than 2 times ULN (3 times ULN for liver metastases)

Renal:

* Creatinine less than 2.2 mg/dL
* NCI renal toxicity no greater than grade 2
* No hypercalcemia (antihypercalcemic therapy allowed)

Cardiovascular:

* Ejection fraction at least 45% by MUGA
* No abnormal ECG or MUGA
* No myocardial infarction within the past year

Pulmonary:

* No abnormal chest x-ray
* FEV_1 greater than 50% of predicted

Other:

* No known allergy to ingredients of study drug
* No known allergy to Staphylococcus aureus Protein A
* HIV negative
* No chronic medical or psychiatric condition that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 30 days since prior biologic therapy (e.g., antibodies, cytokines, or co-stimulatory pathway inhibitors)
* No other concurrent biologic therapy

Chemotherapy:

* See Disease Characteristics
* At least 6 weeks since prior chemotherapy and recovered
* No prior chemotherapy for RCC
* No prior anthracyclines
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* Concurrent steroids allowed
* Concurrent hormonal therapy allowed

Radiotherapy:

* See Disease Characteristics
* No prior mediastinal radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from any recent prior surgery

Other:

* At least 30 days since prior investigational drug or device
* At least 30 days since prior systemic therapy
* No other concurrent investigational drugs
* No other concurrent systemic agents or cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04; Primary Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arie Belldegrun, MD, FACS, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania